CLINICAL TRIAL: NCT02697552
Title: A Phase 1 Open-label Dose Escalation Study to Evaluate the Safety and Pharmacokinetics of HBI-8000 in Japanese Patients With Non Hodgkin's Lymphoma
Brief Title: Safety Study of HBI-8000 in Japanese Patients With Non Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HUYABIO International, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBI-8000-201
Record Dates: First submitted 2016-02-17; First posted 2016-03-03 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — HBI-8000; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HBI-8000 (Experimental): HBI-8000 at the assigned dose twice weekly.
  Interventions: Drug: HBI-8000

INTERVENTIONS:
Drug: HBI-8000 — Oral doses of 30mg, 40mg, 50mg twice weekly [BIW].
  Other Names: Chidamide, CS055

SUMMARY:
Phase 1, open-label, non-randomized, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of HBI-8000 administered orally.

DETAILED DESCRIPTION:
Phase 1, open-label, non-randomized, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary efficacy of HBI-8000 administered orally. Patients must be hospitalized as per guidance of the treating investigator throughout Cycle 1. Patients will receive HBI 8000 twice weekly (BIW) (after breakfast), in 28 day treatment cycles.

Patients will be enrolled in cohorts of 3 patients. The first cohort of 3 patients will receive 30 mg BIW. Decisions regarding cohort escalation will be based upon the clinical experience in Cycle 1 (first 28 days) only. For a given cohort, if 1 patient enrolled in the cohort experiences a dose limiting toxicity (DLT) within 28 days of the first dose, the cohort will be expanded to 6 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically diagnosed non Hodgkin's lymphoma patients for whom no other standard therapy is available
2. Male or female, aged 20 years or over at time of signing informed consent
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 and life expectancy, per the investigator, of more than 3 months at time of signing informed consent
4. Patients for whom at least 1 measurable lesion is confirmed in the lesion assessment before the start of study drug administration
5. Patients must have recovered to Grade 1 or less (Common Terminology Criteria for Adverse Events [CTCAE], Version 4.03) from all toxicity associated with previous chemotherapy, antibody, or radiotherapy. (Exception: patients may enter with continuing alopecia regardless of CTCAE grade.) The following intervals between ending of another treatment and starting of HBI-8000 must elapse:

   * Chemotherapy: 4 weeks
   * Nitrosourea: 6 weeks
   * Radiotherapy: 4 weeks
   * Major surgery: 4 weeks
   * Immunomodulatory drugs: 4 weeks
   * Any antibody agent: 12 weeks (84 days)
   * Autologous stem cell transplantation (ASCT): 12 weeks (84 days)
6. Patients must agree not to consume grapefruit, grapefruit juices, Seville oranges, St.John's wort, or any products containing Seville oranges, grapefruit, or St. John's wort during their participation on the study
7. Patients who signed the informed consent form and are capable of giving informed consent in accordance with the policies of the Institutional Review Board (IRB)
8. Patients must be willing to be hospitalized as per guidance of the treating investigator throughout Cycle 1

Exclusion Criteria:

1. Patients with current, previous, or clinically suspected invasion of the central nervous system (CNS)
2. Organ transplant recipients
3. Allogeneic stem cell transplant recipients
4. Previous extensive radiotherapy involving ≥30% of hematopoietic bone marrow, excluding patients who have had total body irradiation as part of a conditioning regimen for ASCT
5. Patients with an electrocardiogram (ECG) finding at screening of QT interval corrected for heart rate using Fridericia's method (QTcF) prolongation >450 ms in male patients and >470 ms in female patients, ventricular tachycardia, ventricular fibrillation, second- or third-degree heart block, unstable angina, coronary angioplasty or stenting, myocardial infarction, chronic congestive heart failure (New York Heart Association Class III or IV) within 6 months of starting the study drug, any cardiomyopathy, or long QT syndrome
6. Any condition including the presence of laboratory abnormalities, which, as judged by the investigator, places the patient at unacceptable risk if he/she were to participate in the study. Examples of such medical conditions are, but are not limited to, as follows:

   • Uncontrolled diabetes mellitus (e.g., glycosylated hemoglobin [HbA1c] >8%), as judged by the investigator
7. Patients who have had any of the following abnormal measurements at screening performed within 2 weeks (14 days) prior to the start of study drug administration:

   * Hemoglobin: <8 g/dL
   * Neutrophil count: <1,200/µL
   * Platelet count: <75,000/µL
   * Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT): >3 x the upper limit of normal (ULN)
   * Bilirubin level: >1.5 x ULN
   * Creatinine clearance: <50 mL/min via Cockcroft-Gault formula ; proteinuria > Grade 2
   * Plasma troponin I (or troponin T): >ULN
   * Prothrombin time or activated partial thromboplastin time: >1.25 x ULN
   * Potassium, corrected calcium , or magnesium levels outside normal limits
8. Any cardiac arrhythmia requiring anti-arrhythmic medication
9. Patients with a history of seizures
10. Patients with known hypersensitivity to histone deacetylase (HDAC) inhibitors or any of the components of the HBI-8000 tablets
11. Patients with a history or complication of malignant tumors, unless the patients have been free of the disease for 5 years or longer, except the following, if successfully treated, in which case they are not excluded:

    * Basal cell carcinoma of the skin
    * Squamous cell carcinoma of the skin
    * Cervical carcinoma in situ
    * Carcinoma in situ of the breast
    * An incidental histological finding of prostate carcinoma (TNM stage T1a or T1b)
    * Early-stage gastric cancer treated with endoscopic mucosal resection or endoscopic submucosal dissection
12. Patients with uncontrolled inter-current infection
13. Patients with active clinically significant bleeding or recently occurred thrombotic diseases, including patients who are at a high risk for a thromboembolic event and are not willing to take venous thromboembolic prophylaxis
14. Women who are pregnant, women who are not willing to stop breastfeeding during study period and for 10 days after the last dose of study drug, women of child bearing potential, or men with a sexual partner of child bearing potential who are not willing to use double-barrier method during study period and at least 3 months (for men) or at least 1 month (for women) after the last dose of study drug. Double-barrier method is defined as a combination of 2 effective contraceptive methods, such as condom or condom containing spermicide in combination with a diaphragm, oral contraceptive, or intrauterine device.

    Note: Female subjects will be considered to be a woman of childbearing potential unless having undergone permanent contraception or postmenopausal. Postmenopausal is defined as at least 12 months without menses with no other medical reasons (i.e., chemical menopause because of treatment with anti-malignant tumor agents).
15. Seropositivity for the human immunodeficiency virus (HIV) antibody
16. Hepatitis B surface antigen-positive, or hepatitis C virus antibody positive. In case hepatitis B core antibody and/or hepatitis B surface antibody is positive even if hepatitis B surface antigen negative, a hepatitis B virus deoxyribonucleic acid (DNA) test [real-time polymerase chain reaction (PCR]) measurement] should be performed and if positive, the patient should be excluded
17. Patients who were in other experimental clinical studies with investigational agents within 30 days before the start of study drug administration (12 weeks for any investigational antibody therapy or investigational ASCT), or in current clinical studies with investigational agents
18. Patients with a history of drug abuse or long-term excessive alcohol consumption which could affect study result assessment
19. Patients considered by the investigator to be unsuitable for the study because of any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from participating in the study, or because of any condition that confounds the ability to interpret data from the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of HBI-8000 in adult Japanese patients with non Hodgkin's lymphoma (NHL) for whom no other standard therapy is suitable based on the frequency of dose-limiting toxicities (DLTs) which occur within 28 days. | 28 days

SECONDARY OUTCOMES:
Pharmacokinetic parameter: area under the plasma concentration-time curve (AUC) measurement at 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 6, 12, 24, 48, and 72 hours. | 28 days
  Plasma concentration of HBI-8000 will be measured following single dose (Days 1-4) and multiple dose (Days 25-28) administration
Pharmacokinetic parameter: maximum observed plasma concentration (Cmax) measurement at 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 6, 12, 24, 48, and 72 hours. | 28 days
  Plasma concentration of HBI-8000 will be measured following single dose (Days 1-4) and multiple dose (Days 25-28) administration
Pharmacokinetic parameter: time of maximum observed plasma concentration (Tmax) at 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 6, 12, 24, 48, and 72 hours. | 28 days
  Plasma concentration of HBI-8000 will be measured following single dose (Days 1-4) and multiple dose (Days 25-28) administration
Pharmacokinetic parameter: apparent terminal half-life (T1/2) at 0.5, 0.75, 1, 1.5, 2, 2.5, 4, 6, 12, 24, 48, and 72 hours. | 28 days
  Plasma concentration of HBI-8000 will be measured following single dose (Days 1-4) and multiple dose (Days 25-28) administration
Anti-tumor activity of HBI-8000 by overall response status based on Cheson's response criteria for NHL and Japan Clinical Oncology Group (JCOG) response criteria for Adult T-Cell Lymphoma (ATL) | Through study completion, an average of 24 weeks.
Safety of HBI-8000 in Japanese patients with NHL for whom no other standard therapy is suitable with incidence and severity of adverse events graded according to the NCI-CTCAE version 4.03 | Through study completion, an average of 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Kensei Tobinai, MD, Principal Investigator — National Cancer Center Hospital Tokyo, Japan
Locations (8):
- Japan (8):
  - Nagoya City University Hospital, Aichi
  - Fukuoka University Hospital, Fukuoka
  - NHO Kyushu Cancer Center, Fukuoka
  - Kagoshima University Medical and Dental Hospital, Kagoshima
  - Tokai University Hospital, Kanagawa
  - NHO Kumamoto Medical Center, Kumamoto
  - NHO Nagasaki Medical Center, Nagasaki
  - National Cancer Center Hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No